CLINICAL TRIAL: NCT02014350
Title: Outcomes Following Delta Xtend Reverse Shoulder System
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: RI2013
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Reverse Total Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- DePuy Delta Xtend RTSA
  Interventions: Device: DePuy Delta Xtend Reverse TSA

INTERVENTIONS:
Device: DePuy Delta Xtend Reverse TSA

SUMMARY:
To collect medium to long-term survivorship implant outcomes on the DePuy Delta Xtend Reverse Shoulder Stystem.

ELIGIBILITY:
Inclusion Criteria:

Patients whom were implanted with the DePuy Delta Xtend Reverse Total Shoulder System in the time frame indicated. Patients must be willing to sign the consent form and complete all follow-up visits.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who were implanted with the DePuy Delta Xtend Reverse Total Shoulder Arthoplasty between 2008-2012
Sampling Method: Probability Sample
Dates: Primary Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 10 years post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States